CLINICAL TRIAL: NCT04615845
Title: An Open Label, Single-center, Phase 1 Study to Evaluate the Safety of Cancer Immunotherapy With Autologous Dendritic Cells in Patients With Metastatic Castration Resistant Prostate Cancer (mCRPC)
Brief Title: Safety Evaluation of Autologous Dendritic Cell Anticancer Immune Cell Therapy (Cellgram-DC-PC)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Difficult recruitment
Sponsor: Pharmicell Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PMC-DC-01
Record Dates: First submitted 2020-10-22; First posted 2020-11-04 (Actual); Last update posted 2023-01-03 (Actual); Status verified 2022-12

CONDITIONS: Castration Resistant Prostate Cancer, CRPC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cellgram-DC-PC (Experimental): Cellgram-DC-PC is injected subcutaneously near the inguinal lymph nodes
  Interventions: Biological: Cellgram-DC-PC

INTERVENTIONS:
Biological: Cellgram-DC-PC — Patients will receive 3 times every 2 weeks injection of Cellgram-DC-PC(Autologous dendritic cell) subcutaneously near the inguinal lymph nodes
  Other Names: Autologous dendritic cell anti-cancer immune cell therapy for prostate cancer treatment

SUMMARY:
This Phase 1 study to evaluate the safety of cancer immunotherapy with autologous dendritic cells(DC) in patients with metastatic castration resistant prostate cancer (mCRPC)

DETAILED DESCRIPTION:
To evaluate the safety of an autologous dendritic cell anticancer immune cell therapy (Cellgram-DC-PC) for the treatment of prostate cancer in patients with metastatic castration-resistant prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. 19 and under 80 years
2. Histologically confirmed prostate adenocarcinoma
3. Patients with stage M1a or M1b with extrapelvic lymph nodes and bone metastases
4. Patients diagnosed with castration-resistant prostate cancer after failure of male hormone deprivation therapy (Castrate levels of testosterone <50 ng/dL) and If either a or b is satisfied:

   1. Biochemical progression: Prostate Specific Antigen (PSA) increases three times in a row at 1 week intervals, two 50% increases compared to the lowest point, PSA> 2ng/mL, or
   2. Radiological progression: appearance of new lesions; 2 or more new lesions on the bone scan
5. Asymptomatic or mild patients after previous treatment

   1. Patients who have not used narcotic analgesics within 21 days prior to enrollment
   2. Patients with an average weekly pain of less than 4 on the Visual Analogue Scale(VAS) (out of 10)
6. Combination of Luteinizing hormone-releasing hormone(LHRH) analogs (leuprolide (Lupron, Viadur, Eligard) and goserelin (Zoladex, etc.) for the inhibition of gonadotropin is allowed
7. Whole body performance status: European Cooperative Oncology Group(ECOG) 0~1
8. Patients whose life expectancy is at least 6 months or longer
9. Hb ≥ 8.0g/dL, Absolute Neutrophil Count(ANC) ≥ 1,500/mm3, Platelets ≥ 100,000/mm3
10. Serum Creatinine ≤ 2.0 x Upper Limit of Normal(ULN) or Calculated Creatinine Clearance > 30mL/min
11. Total Bilirubin ≤ 1.5 x ULN or Direct bilirubin ≤ ULN, Aminotransferase (AST)/Alanine aminotransferase(ALT) <2.5 x ULN
12. Patients who did not receive surgery, radiation therapy, or immunotherapy within the last 6 weeks and recovered from side effects
13. Patients who agreed to use medically recognized contraceptive methods during the clinical trial participation period
14. Patients who voluntarily participated in clinical trials and signed the Informed Contents Form (ICF)

Exclusion Criteria:

1. Patients who have a local recurrence and are scheduled for local treatment.
2. Patients with malignant tumors other than non-melanoma skin cancer in the past 3 years
3. Patients with visceral metastases (metastases to the lungs, liver, adrenal glands, peritoneum, brain, etc.)
4. Patients who previously received anti-tumor immunotherapy (anti-PD1, anti-PDL1 or anti-PDL2, etc.) or participated in immunotherapy-related clinical trials
5. Patients with active autoimmune diseases requiring systemic immunosuppression treatment (e.g., immunosuppressants such as cyclosporin A or azathioprine or steroids for disease control)
6. Patients with medical conditions requiring continuous or intermittent administration of systemic steroids or immunosuppressants
7. Patients who received blood products (limited to whole blood products) within 4 weeks of screening criteria, or patients who received colony stimulating factors (Colony Stimulating Factor or recombinant Erythropoietin)
8. Patients with a history of organ or hematopoietic stem cell transplantation
9. Patients with acute or chronic infections requiring systemic treatment
10. Patients known to be infected with human immunodeficiency virus (HIV)/serum positive
11. Patients with active hepatitis A, B or C
12. Patients with untreated syphilis (Fluorescent Treponemal Antibody Absorption Test (FTA-ABS) Immunoglobulin M positive patients)
13. Patients expected to require therapeutic biotherapy or immunotherapy
14. Patients who received live virus vaccines (e.g. measles, mumps, rubella, chickenpox, yellow fever, rabies, Bacillus Calmette-Guerin (BCG), oral typhoid vaccine, Flu-Mist, etc.) within 30 days
15. Patients with a history of anaphylaxis to gentamicin
16. Others, if the person in charge of the study determines that it is not suitable for the clinical trial

Ages: 19 Years to 79 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
The Measure CTCAE of Safety | For 28 weeks
  The level of Adverse Event (AE) is described in accordance with the Common Terminology Criteria for Adverse Event (CTCAE) (Version 5.0).

SECONDARY OUTCOMES:
Immune response evaluation (INF-r) | 0, 2, 8, 16 and 28 weeks
  The tumor antigen-specific immune response induced after administration compared to before Investigational Product(IP) administration was confirmed by measuring changes in the secretion of cytokines INF-r in serum (ELISA).
Immune response evaluation (IL-12) | 0, 2, 8, 16 and 28 weeks
  The tumor antigen-specific immune response induced after administration compared to before Investigational Product(IP) administration was confirmed by measuring changes in the secretion of cytokines IL-12 in serum (ELISA).
Measurement of changes in tumor marker test results (PSA) | 0, 2, 4, 8, 16 and 28 weeks
  Changes in tumor marker test results (PSA) are measured at each time point (V4, V5, V6, V7, V8) after administration compared to before (V3) Investigational Product(IP) administration.

CONTACTS AND LOCATIONS:
Overall Officials: BUMJIN LIM, Ph.D, Principal Investigator — Asan Medical Center
Locations (1):
- Asan medical center, Seoul, South Korea